CLINICAL TRIAL: NCT04034121
Title: Non-randomized Evaluation of the DESolve® Novolimus Eluting Bioresorbable Coronary Scaffold System in de Novo Native Coronary Artery Lesions - DESolve Cx Single-Arm Registry
Brief Title: Elixir Medical Evaluation of the DESolve® Novolimus Eluting Bioresorbable Coronary Scaffold System - Cx Registry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELX-CL-1003 Cx
Record Dates: First submitted 2019-02-06; First posted 2019-07-26 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Coronary Artery Disease
Keywords: biorersorbable scaffold; drug eluting; novolimus
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- DESolve Cx (Other): DESolve Cx Novolimus Eluting Bioresorbable Coronary Scaffold System
  Interventions: Device: DESolve Cx drug eluting coronary scaffold system

INTERVENTIONS:
Device: DESolve Cx drug eluting coronary scaffold system — percutaneous coronary intervention

SUMMARY:
This additional arm of the DESolve Nx study is an evaluation of the CE Mark approved DESolve Cx Novolimus Eluting Bioresorbable Scaffold System.

DETAILED DESCRIPTION:
The DESolve Cx Single-Arm Registry enrolled patients using the same inclusion and exclusion criteria and clinical endpoints as the DESolve Nx Study

This study was split into 2 cohorts - European and Brazilian. The European cohort (30 subjects) completed all follow-up at 1 year and the Brazilian cohort at 3 years (20 subjects)

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age and for the 35-patient subset, patients must be over the age of 50
* Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the DESolve Novolimus Eluting Bioresorbable Coronary Scaffold System (BCSS) and he/she provides written informed consent, as approved by the appropriate Ethics Committee of the respective clinical site, prior to any clinical study related procedure
* Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or electrocardiogram (ECG) changes consistent with ischemia)
* Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
* Patient must agree to undergo all clinical study required follow-up visits, angiograms, and as applicable, imaging testing
* Patient must agree not to participate in any other clinical study for a period of two years following the index procedure
* Target lesion must be located in a native coronary artery with a nominal vessel
* Not part of a clinical investigation
* Treatment of a single, non-target lesion located in a separate major epicardial vessel Target vessel diameter must be a diameter of between 2.25 and 3.5 mm assessed by online QCA
* Target lesion must measure ≤ 24 mm in length
* Target lesion must be in a major artery or branch with a visually estimated stenosis of ≥ 50% and < 90% with a TIMI flow of ≥ 1
* Target vessel must be in a major coronary artery or major branch

Exclusion Criteria:

* Patient has a known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure and cardiac enzymes have not returned within normal limits at the time of procedure
* Patient is currently experiencing clinical symptoms consistent with AMI
* Patient requires the use of any rotablator intervention during the index procedure
* Patient has current unstable arrhythmias
* Patient has a known left ventricular ejection fraction (LVEF) < 30%
* Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
* Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure
* Patient is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.)
* Patient is receiving chronic anticoagulation therapy (e.g., heparin, coumadin) that cannot be stopped and restarted according to local hospital standard procedures.
* Patient has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, both clopidogrel and ticlopidine, Novolimus, PLLA polymers or contrast sensitivity that cannot be adequately pre-medicated
* Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin or clopidogrel
* Patient has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented or suspected liver disease.
* Patient has known renal insufficiency (e.g., serum creatinine level of more than 2.5 mg/dL, or patient on dialysis)
* Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
* Patient has had a significant GI or urinary bleed within the past six months
* Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion
* Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical study plan, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year)
* Patient is already participating in another clinical study
* Women of childbearing potential who have not undergone surgical sterilization or are not post-menopausal (defined as amenorrheic for at least one year) as well as women who are pregnant or nursing
* Patient is unable to give their consent, is legally incompetent, or is institutionalized by virtue of an order issued by the courts or other authority
* Target lesion(s) meets any of the following criteria:
* Aorto-ostial location
* Left main location
* Located within 5 mm of the origin of the LAD or LCX
* Located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft
* Lesion involving a side branch >2mm in diameter or bifurcation
* Previous placement of a scaffold proximal to or within 10 mm of the target lesion
* Total occlusion (TIMI flow 0), or TIMI flow < 1
* Excessive tortuosity proximal to or within the lesion
* Angulation (≥ 45o) proximal to or within the lesion
* Calcification moderate or heavy
* Previous intervention restenosis
* The target vessel contains visible thrombus
* Another clinically significant lesion (>40%) is located in the same major epicardial vessel as the target lesion
* Patient has a high probability that a procedure other than pre-dilatation and scaffolding and (if necessary) post-dilatation will be required at the time of index procedure for treatment of the target vessel (e.g. atherectomy, cutting balloon or brachytherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2017-01-22 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Verheye, MD, Principal Investigator — ZNA Antwerp Belgium
Locations (3):
- Belgium (2):
  - AZ Middelheim Hospital, Antwerp
  - St. - Jan Ziekenhuis Z.O.L., Genk
- Instituto Dante Pazzanese, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 20 January 2016 and 18 July 2016 Nov 2017, 50 patients were enrolled in the study at 3 centers in Brazil (20 patients) and Belgium (30 patients)
Groups:
- DESolve Cx: DESolve Cx Novolimus Eluting Bioresorbable Coronary Scaffold System
  The DESolve Cx Novolimus Eluting BCSS is comprised of four main components: the Poly-L-Lactic Acid-based polymer (PLLA) stent coated with a PLLA-based polymer-drug matrix containing the anti-proliferative drug Novolimus.
Period: European Cohort
Arm/Group | DESolve Cx
Started | 30 (The European Cohort enrolled 30 patients)
Completed | 30
Not Completed | 0
Period: Brazil Cohort
Arm/Group | DESolve Cx
Started (20 patients enrolled in Brazil continued follow-up through 3 years) | 20 (The Brazil Cohort enrolled 20 patients)
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DESolve Cx
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 60.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 30
  Brazil | 20
Cardiac Risk Factors [Count of Participants; unit: Participants] — The same participant may be included in more than one category therefore the number of participants does not equal the total number of participants in the group.
  Participants
    Diabetes | 10
    Hypertension | 35
    Dyslipidemia | 42
    Family history of coronary artery disease | 24
    Smoking (previous or current) | 35
    Prior myocardial infarction | 20
    Prior percutaneous coronary intervention | 13
Baseline Lesion Characteristics [Mean (Standard Deviation); unit: mm]
  Reference Vessel Diameter | 3.03 (0.39)
  Minimum Lumen Diameter | 1.17 (0.30)
  Lesion Length | 16.16 (6.55)
Percent Diameter Stenosis [Mean (Standard Deviation); unit: Percent] | 61.20 (9.27)

OUTCOME MEASURES:

1. Primary Outcome: Clinically-indicated Major Adverse Cardiac Events
Description: Number of Participants with one or more Clinically-indicated Major Adverse Cardiac Events This applies to the European and Brazilian Cohorts
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | DESolve Cx
Number analyzed (Participants) | 50
Participants | 0

2. Secondary Outcome: In-scaffold Late Lumen Loss by Quantitative Coronary Angiography (QCA)
Description: quantitative QCA measurement of change in the lumen diameter from post procedure and 6 months which is described as "late lumen loss" This applies to both the European and Brazilian Cohorts
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | DESolve Cx
Number analyzed (Participants) | 50
mm | 0.19 (0.25)

3. Secondary Outcome: Clinically-indicated Major Adverse Cardiac Events (MACE)
Description: Number of Participants with one or more Clinically-indicated Major Adverse Cardiac Events This applies to both the European and Brazilian Cohorts
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | DESolve Cx
Number analyzed (Participants) | 50
Participants | 0

4. Secondary Outcome: Clinically-Indicated Major Adverse Cardiac Events
Description: Number of Participants with one or more Clinically-indicated Major Adverse Cardiac Events This time point applies to the Brazilian Cohort only
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | DESolve Cx
Number analyzed (Participants) | 20
Participants | 0

5. Secondary Outcome: Clinically-indicated Major Adverse Cardiac Events
Description: Number of Participants with one or more Clinically-indicated Major Adverse Cardiac Events This applies to the Brazilian Cohort only
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | DESolve Cx
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: Major Adverse Event data was collected at 1 month, 6 months, 1, 2 and 3 years. MACE was defined as a composite endpoint of cardiac death, target vessel MI, and clinically-indicated target lesion revascularization.
Arm/Group | DESolve Cx
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DESolve Cx (N=50)
non-clinically indicated target lesion revascularization (Cardiac disorders) | 2 (2) — Revascularization of the target lesion not meeting the definition of clinically-indicated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: European Cohort (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT04034121/Prot_000.pdf
  • Study Protocol: Brazil Cohort (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT04034121/Prot_001.pdf
  • Informed Consent Form: European Cohort (2015-10-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT04034121/ICF_002.pdf